CLINICAL TRIAL: NCT06589765
Title: A Phase 3, Randomized, Double-blinded Study to Evaluate the Efficacy and Safety of HRS-7535 Compared With Dapagliflozin in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Metformin (OUTSTAND-2)
Brief Title: A Study of HRS-7535 Compared With Dapagliflozin in Adult Participants With Type 2 Diabetes and Inadequately Controlled With Metformin
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRS-7535-302
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: HRS-7535 tablet compared with dapagliflozin tablet
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Experimental): subjects will receive HRS-7535 tablet orally at dose 1.
  Interventions: Drug: HRS-7535 tablet
- Treatment group B (Experimental): subjects will receive HRS-7535 tablet orally at dose 2.
  Interventions: Drug: HRS-7535 tablet
- Treatment group C (Experimental): subjects will receive HRS-7535 tablet orally at dose 3.
  Interventions: Drug: HRS-7535 tablet
- Treatment group D (Active Comparator): subjects will receive dapagliflozin tablet orally.
  Interventions: Drug: dapagliflozin tablet

INTERVENTIONS:
Drug: HRS-7535 tablet — HRS-7535 tablet
  Arms: Treatment group A; Treatment group B; Treatment group C
Drug: dapagliflozin tablet — dapagliflozin tablet
  Arms: Treatment group D

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of HRS-7535 compared with dapagliflozin in subjects with type 2 diabetes mellitus with inadequate glycemic control using metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 age years, both inclusive;
2. Type 2 diabetes mellitus diagnosed for at least 3 months before the screening visit;
3. HbA1c 7.5-11.0% (both inclusive) at screening;
4. Treated with conventional lifestyle intervention and stable treatment with metformin (≥1500 mg/day) at least 8 weeks prior to screening.

Exclusion Criteria:

1. Known or suspected allergy to the investigational drug or its components or excipients.
2. Diagnosed or suspected with type 1 diabetes mellitus, special types of diabetes or secondary diabetes.
3. Have a history of acute complications of diabetes (diabetic ketoacidosis, lactic acidosis, hyperglycaemic hyperosmolar state, etc.) within 6 months prior to screening.
4. Proliferative retinopathy, maculopathy, painful diabetic neuropathy, diabetic foot ulcer or intermittent claudication requiring acute treatment;
5. Pregnancy, breast-feeding, intention of becoming pregnant during the trial; or women of childbearing potential (WOCBP) or male subject not using adequate contraceptive measures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 32 weeks of treatment | at 32 weeks

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved HbA1c <7.0% at Week 32 | at 32 weeks
Percentage of Participants Who Achieved HbA1c ≤6.5% at Week 32 | at 32 weeks
Change from Baseline in Fasting Serum Glucose, from Baseline to Week 32 | at 32 weeks
Percentage Change from Baseline in Body Weight, from Baseline to Week 32 | at 32 weeks
Change from Baseline in Body Weight, from Baseline to Week 32 | at 32 weeks
Change from Baseline in Waist Circumference, from Baseline to Week 32 | at 32 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided